CLINICAL TRIAL: NCT05235880
Title: Effects of Virtual Reality Based Games on Upper Extremities, Trunk and Cognitive Functions in Parkinson's Disease
Brief Title: Effects of Virtual Reality Based Games in Rehabilitation of Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Muhammed KILINÇ, Associate Professor, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KA-21067
Record Dates: First submitted 2021-12-22; First posted 2022-02-11 (Actual); Last update posted 2023-09-21 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: parkinson disease; physiotherapy; exergames
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): 1 hour physiotherapy session for 3 times a week and 8 weeks in total.
  Interventions: Other: Virtual reality based games
- control group (Active Comparator): 1 hour physiotherapy session for 3 times a week and 8 weeks in total.
  Interventions: Other: Conventional exercises

INTERVENTIONS:
Other: Virtual reality based games — In an hour physiotherapy session first 40 minutes of session includes conventional physiotherapy program tailored to patient's needs. Last 20 minutes of session includes virtual reality based games aiming improvement on upper extremities, trunk and cognitive functions.
  Arms: study group
Other: Conventional exercises — In an hour physiotherapy session first 40 minutes of session includes conventional physiotherapy program tailored to patient's needs. Last 20 minutes of session includes conventional physiotherapy approaches aiming improvement on upper extremities, trunk and cognitive functions.
  Arms: control group

SUMMARY:
The purpose of this study is to investigate the effects of virtual reality based games on upper extremities, trunk and cognitive functions in patients with Parkinson's Disease.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Parkinson's disease
* 50 years old and over
* Stage 1.5-3 according to the modified Hoehn-Yahr Staging Scale
* Mini mental test score of 24 and above

Exclusion Criteria:

* Additional neurological disease or symptom other than Parkinson's disease
* Orthopedic disorder that will prevent them from doing exercises
* Severe mental disorders

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-15 (Actual); Primary Completion 2023-06-15 (Actual); Study Completion 2023-06-15 (Actual)

PRIMARY OUTCOMES:
Upper extremities performance with 9 hole peg test | Change from Baseline at 8 weeks
  The patient sits with a table in front of him/her and places 9 small wooden sticks on the surface with nine holes on them, takes them out again and lays them on his/her side. He/she is asked to do it as quickly as possible and his/her time is saved
Upper extremities performance with Minnesota Manual Dexterity Test | Change from Baseline at 8 weeks
  It involves taking small disc-shaped objects, each of standard size, to different distances on the table in the shortest possible time and placing them in sequence, while the patient is in a sitting position with a table in front of him/her.
Cognitive Status with Montreal Cognitive Assessment | Change from Baseline at 8 weeks
  its validity and reliability in Turkish have been established. The total score ranges from 0-30, and a higher score indicates a better cognitive status. Below 21 points indicates cognitive impairment.
Trunk Functions with Trunk Impairment Scale | Change from Baseline at 8 weeks
  It is a valid and reliable scale for evaluating the motor disorders and balance of the trunk in Parkinson's patients. The total score in the scale, which consists of 17 items in 3 sections, ranges from 0 to 23. A higher score indicates better trunk function and balance.

SECONDARY OUTCOMES:
Dynamic balance with functional reach test | Change from Baseline at 8 weeks
  Functional reach test is frequently used to assess dynamic balance and fall risk. While the patient is standing by the wall, he/she raises his/her arm to 90 degrees and tries to reach as far as he/she can without taking his/her feet off the ground. Extending a longer distance indicates better balance and less risk of falling
Balance and mobility with Timed Up and Go Test | Change from Baseline at 8 weeks
  While the patient is in a sitting position, he/she is asked to stand up from the chair, walk 3 meters, turn around, come back and sit down, and the time is recorded. Doing it in less time demonstrates better balance and mobility
Quality of life with Parkinson's Disease Questionnaire | Change from Baseline at 8 weeks
  The 39-item Parkinson's Disease Questionnaire was developed to evaluate the quality of life of Parkinson's patients and has Turkish validity and reliability. Higher scores mean worse outcome.
Disease severity and symptoms with Unified Parkinson Disease Rating Scale Part 2 and 3 | Change from Baseline at 8 weeks
  It is one of the most frequently used scales to evaluate the severity of the disease in Parkinson's patients. It evaluates many problems such as motor and non-motor problems, treatment complications, problems in daily living activities and consists of 4 sections. However, in our study, the 2nd and 3rd sections which evaluate motor problems and activities of daily living will be used. Higher scores mean worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Gül Yalçın Çakmaklı, Assoc. Prof., Principal Investigator — Hacettepe University
Locations (1):
- Hacettepe University, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kalia LV, Lang AE. Parkinson's disease. Lancet. 2015 Aug 29;386(9996):896-912. doi: 10.1016/S0140-6736(14)61393-3. Epub 2015 Apr 19. PMID 25904081
- [Background] Jankovic J. Parkinson's disease: clinical features and diagnosis. J Neurol Neurosurg Psychiatry. 2008 Apr;79(4):368-76. doi: 10.1136/jnnp.2007.131045. PMID 18344392
- [Background] Abbruzzese G, Marchese R, Avanzino L, Pelosin E. Rehabilitation for Parkinson's disease: Current outlook and future challenges. Parkinsonism Relat Disord. 2016 Jan;22 Suppl 1:S60-4. doi: 10.1016/j.parkreldis.2015.09.005. Epub 2015 Sep 3. PMID 26360239
- [Background] Allen NE, Song J, Paul SS, Smith S, O'Duffy J, Schmidt M, Love R, Sherrington C, Canning CG. An interactive videogame for arm and hand exercise in people with Parkinson's disease: A randomized controlled trial. Parkinsonism Relat Disord. 2017 Aug;41:66-72. doi: 10.1016/j.parkreldis.2017.05.011. Epub 2017 May 15. PMID 28528804
- [Background] Levin MF. Can virtual reality offer enriched environments for rehabilitation? Expert Rev Neurother. 2011 Feb;11(2):153-5. doi: 10.1586/ern.10.201. No abstract available. PMID 21306202
- [Derived] Cetin B, Kilinc M, Cakmakli GY. The effects of exergames on upper extremity performance, trunk mobility, gait, balance, and cognition in Parkinson's disease: a randomized controlled study. Acta Neurol Belg. 2024 Jun;124(3):853-863. doi: 10.1007/s13760-023-02451-3. Epub 2024 Jan 5. PMID 38182919